CLINICAL TRIAL: NCT01079663
Title: The Efficacy and Safety of Chlorhexidine Gluconate Chip (Periochip®) in Therapy of Symptoms in Patients With Peri-implantitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI/013P
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chlorhexidine chip (Periochip®) (Experimental): PerioChip®, consisting of 2.5 mg Chlorhexidine Gluconate PerioChips were inserted only to target pockets whose pocket depth (PD) at Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 12 and Week 18 was ≥ 6 mm
  Interventions: Drug: Chlorhexidine 2.5 mg
- Placebo chip (Placebo Comparator): Placebo Chip Placebo Chips were inserted only to target pockets whose pocket depth (PD) at Baseline visit (Week 0), Week 2, Week 4, Week 6, Week 8, Week 12 and Week 18 was ≥ 6 mm
  Interventions: Drug: Placebo chip

INTERVENTIONS:
Drug: Chlorhexidine 2.5 mg
  Arms: Chlorhexidine chip (Periochip®)
Drug: Placebo chip
  Arms: Placebo chip

SUMMARY:
The purpose of the study is to assess the efficacy and the safety of Chlorhexidine Gluconate chip (Periochip®) versus Placebo Chip in treatment of symptoms in patients with Peri-Implantitis.

DETAILED DESCRIPTION:
This is a Phase 2a study assessing the safety and efficacy of Chlorhexidine Gluconate chip (Periochip®) versus Placebo Chip in treatment of symptoms in patients with Peri-Implantitis

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form.
2. Good general health.
3. Male or female patients aged >21 years old.
4. Availability for the 25 week duration of the study.
5. Peri-implantitis is characterized by the presence of at least 1 implant with periodontal pockets of 6-10 mm in depth (potential target implant) demonstrating Bleeding on Probing without involving the apex of the implant and confirmed radiographically.
6. Females of childbearing potential must be non-pregnant and non-lactating at entry and agree to use an adequate method of birth control during the study.

Exclusion Criteria:

1. Presence of oral local mechanical factors that could (in the opinion of the Investigator) influence the outcome of the study.
2. Presence of orthodontic appliances, or any removable appliances, that impinges on the tissues being assessed.
3. Presence of soft or hard tissue tumours of the oral cavity.
4. Horizontal inter implant distance ≤2 mm (if an adjacent implant exists).
5. Selection of the following dental implant types as target implant/s: hydroxylapatite (HA) and/or Titanium Plasma-sprayed (TPS).
6. History of allergy to Chlorhexidine.
7. Patients treated with systemic antibiotic therapy or periodontal/mechanical/local delivery therapy within 6 weeks prior to study entry and throughout the study duration.
8. Patients treated with non-steroidal anti-inflammatory drugs (NSAIDs) within 14 days prior to entry into the study and throughout the study duration (excluding treatment of acetylsalicylic acid ≤100 mg /day).
9. Patients taking Phenytoin, calcium channel blockers drugs (CCBs) and/or cyclosporine, which might influence the pattern of tissue response.
10. Presence of any of the following conditions: Type 1 diabetes, major recurrent aphtae stomatitis, abscesses and related oral pathologies.
11. The presence of any medical or psychiatric condition or any other condition that, in the opinion of the Investigator, could affect the successful participation of the patient in the study.
12. Patient participates in any other clinical study 30 days prior to the start of the study and throughout the study duration.
13. Patient uses Chlorhexidine oral rinses/ mouthwashes on a regular basis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Periodontology, School of Graduate Dentistry, Rambam Health Care Center, Haifa
  - The Oral & Maxillofacial Surgery Unit of the Tel Aviv Medical Center, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Chlorhexidine Chip (Periochip®): PerioChip®, consisting of 2.5 mg Chlorhexidine Gluconate
  Chlorhexidine 2.5 mg
- Placebo Chip: Placebo chip
Period: Overall Study
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip
Started | 30 | 30
Completed | 30 | 26
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (10.51) | 60.1 (7.88) | 58.4 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 10 | 15 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Israel | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Probing Pocket Depth (PPD) for Selected Target Pocket
Description: Pocket depth is the measurement of the distance from the coronal edge of the gingival margin to the base of the pocket. Measurements were taken with a standard 15-mm University of North Carolina (UNC) periodontal probe.
  Change from baseline in PPD was calculated as Week 24 PPD minus Baseline PPD such that a negative difference indicates an improvement in condition
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target implant
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip
Number analyzed (Participants) | 30 | 30
Number analyzed (Target implant) | 40 | 37
mm | -2.13 (1.399) | -1.79 (1.149)
Statistical Analysis 1: Comparison: Chlorhexidine Chip (Periochip®) vs Placebo Chip; Test type: Superiority; p = 0.1629, Mixed Models Analysis; Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-1.19 to 0.20]

2. Secondary Outcome: Clinical Attachment Levels (CAL)
Description: Loss of attachment is defined as the distance in millimetres that the base of the pocket has migrated apically from the gingival margin of the crown. CAL was calculated at the same site that PPD was measured
Time Frame: Baseline to Week 24
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Target implant
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip
Number analyzed (Participants) | 30 | 30
Number analyzed (Target implant) | 40 | 37
mm | -2.18 (1.394) | -1.76 (1.257)
Statistical Analysis 1: Comparison: Chlorhexidine Chip (Periochip®) vs Placebo Chip; Test type: Superiority; p = 0.0347, Mixed Models Analysis; Mean Difference (Final Values) = -0.76, 95% CI 2-sided [-1.46 to -0.06]

3. Secondary Outcome: Bleeding on Probing (BOP)
Description: BOP was measured at the same site after measuring the PPD. The scoring system used for recording the BOP was a dichotomous one:
  0 = No bleeding
  1 = Bleeding on probing of the pocket base
Time Frame: Baseline to Week 24
Measure: Count of Units; unit: Target implant
Units Other Than Participants: Target implant
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip
Number analyzed (Participants) | 30 | 30
Number analyzed (Target implant) | 40 | 37
Target implant | 23 | 16

ADVERSE EVENTS:
Time Frame: Baseline through Week 24
Description: All patients who receive study drug and have at least one follow-up assessment after beginning treatment
Arm/Group | Chlorhexidine Chip (Periochip®) | Placebo Chip
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 2/30
Other Adverse Events (participants affected / at risk) | 15/30 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine Chip (Periochip®) (N=30) | Placebo Chip (N=30)
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorhexidine Chip (Periochip®) (N=30) | Placebo Chip (N=30)
Aphthous ulcer (Gastrointestinal disorders) | 1 | 2
Gingival swelling (Gastrointestinal disorders) | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 3 | 0
Periodontal inflammation (Gastrointestinal disorders) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 2
Implant site pain (General disorders) | 2 | 4
Feeling cold (General disorders) | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 2
Tooth extraction (Surgical and medical procedures) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No